CLINICAL TRIAL: NCT01672684
Title: At-Home Support for Rural Women Using Group Video Calling
Brief Title: Phase I: At-Home Support for Rural Women Using Group Video Calling
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: California Breast Cancer Research Program (Other)
Responsible Party: Principal Investigator, Cheryl Koopman, Professor (Research) of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BRSADJ0023; NCI-2012-01357 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21349 (Other: Stanford University)
Record Dates: First submitted 2012-08-20; First posted 2012-08-27 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Depression; Post-traumatic Stress Disorder; Recurrent Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
Keywords: quality of life
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic; Breast Neoplasms | interventions — Early Intervention, Educational; Methods

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (experimental arm) (Experimental): Participants complete at-home group video calling sessions for 1 1/2 hours once weekly for 8 weeks.
  Interventions: Procedure: support group therapy
- Arm II (control arm) (Active Comparator): Participants receive an educational workbook journal.
  Interventions: Other: educational intervention

INTERVENTIONS:
Procedure: support group therapy — Complete at-home group video calling support sessions
  Arms: Arm I (experimental arm)
Other: educational intervention — Receive an educational workbook journal
  Other Names: intervention, educational
  Arms: Arm II (control arm)

SUMMARY:
This randomized phase I trial studies at-home group video calling sessions in quality of life in rural patients with breast cancer. At-home group video calling support sessions may improve the well-being and quality of life of women who have breast cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine whether delivering at-home professionally-led breast cancer support using group video calling is feasible, acceptable and satisfactory for women in rural northern California.

II. To evaluate the feasibility of using on-line tools to recruit, screen, treat, and assess this population for a subsequent randomized clinical trial.

III. Assess whether the rate of recruitment of women in this region in this study using predominantly on-line means of recruitment can be improved over that of the previous study using predominantly face-to-face means of recruitment.

SECONDARY OBJECTIVES:

I. Estimate effect size changes in measures of quality of life (post-traumatic stress disorder symptoms, depression symptoms, perceived stress, and positive states of mind), satisfaction with social support, and self-efficacy for coping with cancer.

II. Prescribe sample size. III. Perform I and II for all of these outcomes.

OUTLINE: Participants are randomized to 1 of 2 treatment arms.

ARM I (experimental arm): Participants complete at-home group video calling sessions for 1 1/2 hours once weekly for 8 weeks.

ARM II (control arm): Participants receive an educational workbook journal.

After completion of study treatment, participants are followed up for 1 week.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for this study, the participant must have been diagnosed with breast cancer within the previous 5 years prior to study entry; individuals who have been diagnosed with any stage of breast cancer are eligible
* There are no limitations regarding allowable type and amount of prior therapy
* There are no race/ethnic restrictions
* There are no life expectancy restrictions
* Neither Eastern Cooperative Oncology Group (ECOG) nor Karnofsky performance status will be employed
* There are no requirements for organ and marrow function
* Ability to understand and the willingness to sign a written informed consent document; this will be assessed in the telephone screen conducted by Lisa Frankel as she will review each section of the consent form with the participant and ask if she has any questions about it; this telephone screen will have been approved by the Stanford University Institutional Review Board (IRB), and Lisa Frankel will conduct the interviews in a private location to ensure confidentiality
* Eligibility for this study requires that a woman be a resident of one of 27 rural counties in California (Alpine, Amador, Butte, Calaveras, Colusa, Del Norte, El Dorado, Glenn, Imperial, Inyo, Lake, Lassen, Madera, Mariposa, Modoc, Mono, Nevada, Placer, Plumas, Shasta, Sierra, Siskiyou, Sutter, Tehama, Trinity, Tuolumne, or Yuba, except we will not include women living within the following cities: Chico, Madera, Redding, Rocklin, Roseville or Yuba City, due to this study's more rural focus)
* Eligibility for this study requires that a woman has sufficient hearing to be able to engage in conversation over the phone
* Eligibility for this study requires that a woman has a private place available where she can access the internet
* Eligibility for this study requires that a woman is potentially available to meet at the day of the week and time of the day that the group intervention is scheduled Ã¢ in the event that she is randomly assigned to receive the at-home group calling intervention
* Eligibility for this study requires that women have broadband or digital subscriber line (DSL) internet access
* Eligibility for this study requires that women have a computer with a webcam and either a microphone or a phone available to call into the video conference

Exclusion Criteria:

* There are no therapy restrictions
* There are no restrictions regarding use of other investigational agents
* There are no exclusion requirements due to co-morbid disease or incurrent illness
* Requirements regarding history of allergic reactions attributed to compounds of similar chemical or biologic composition to investigational agent or device are not applicable to this study
* There are no exclusion criteria relating to concomitant medications or substances that have the potential to affect the activity or pharmacokinetics of the study agent
* There are no other agent-specific exclusion criteria
* Pregnancy or nursing patients will not be excluded from the study
* Patients who are cancer survivors or those who are human immunodeficiency virus (HIV)-positive will not be excluded from the study

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of the study protocol as determined primarily through qualitative analysis of the group sessions and the interview data | At 1 week post-intervention
  The major criterion for determining feasibility is to determine whether we can recruit rural women with breast cancer more rapidly using predominantly on-line procedures in this study than in our previous study that predominantly used face-to-face procedures. The qualitative data for determining the feasibility will be collected during the at-home group video calling sessions and from women's interviews conducted at the end of the study. Will be assessed using mixed methods.
Acceptability of the study protocol as determined primarily through qualitative analysis of the group sessions and the interview data | At 1 week post-intervention
  The qualitative data for determining the acceptability will be collected during the at-home group video calling sessions and from women's interviews conducted at the end of the study. Will be assessed using mixed methods.

SECONDARY OUTCOMES:
Changes in quality of life (posttraumatic stress, depression symptoms, perceived stress, and positive states of mind) | From baseline to 1 week post-intervention
  Treatment effect size will be estimated for each measure for the purpose of prescribing the sample size for a subsequent larger randomized clinical trial examining efficacy of the intervention. Will be analyzed using generalized linear mixed models.
Changes in satisfaction with social support | From baseline to 1 week post-intervention
  Treatment effect size will be estimated for each measure for the purpose of prescribing the sample size for a subsequent larger randomized clinical trial examining efficacy of the intervention. Will be analyzed using generalized linear mixed models.
Changes in self-efficacy for coping with cancer | From baseline to 1 week post-intervention
  Treatment effect size will be estimated for each measure for the purpose of prescribing the sample size for a subsequent larger randomized clinical trial examining efficacy of the intervention. Will be analyzed using generalized linear mixed models.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Koopman, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Sierra Streams Institute, Nevada City, California
  - Stanford University Cancer Institute, Stanford, California